CLINICAL TRIAL: NCT00852735
Title: Effect of the Antioxidant Micronutrients of Rapeseed Oil on the Prevention of Cardiovascular Diseases
Brief Title: Effect of the Antioxidant Micronutrients of Rapeseed Oil on the Prevention of Cardiovascular Diseases (Optim'Oils)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); ITERG (Industry); Unilever R&D (Industry); Lesieur (Industry)
Responsible Party: Noël CANO, CRNH Auvergne
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CHU-0047; AU 759
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular diseases; Rapeseed oil; Micronutriments; HDL cholesterol; Oxidative stress; Tocopherols; Sterols; Prevention of cardiovascular diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Rapeseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Dietary Supplement: Rapeseed Oil (prevention of cardiovascular diseases) — to assess the effect of optimized oil (enriched with micronutriments) on the prevention on cardiovascular diseases

SUMMARY:
The purpose of this study is to assess the effect of optimized oil (enriched with micronutriments) on the prevention on cardiovascular diseases.

Randomised crossover dietary intervention study:

The main objective of the clinical study is to investigate the effect of the consumption of an "optimized" rapeseed oil on the lipid metabolism of volunteers as compared with the consumption of a "reference" oil.

Post prandial study:

The second objective of the clinical study is to investigate the effect of the consumption of an "optimized" rapeseed oil on the biomarkers of oxidative stress during post prandial period as compared with the consumption of a "reference" oil.

DETAILED DESCRIPTION:
For both studies, sedentary men between 30 and 65 years of age, with a BMI between 25 and 30, without cardiovascular disorders, will be selected.

Randomised crossover dietary intervention study:

Sixty volunteers will be randomised into 2 groups of 30. The study will last 12weeks. The first 3 weeks will be an adaptation period or "run in". Volunteers will have every day20 g of the reference rapeseed oil and 20 g of the reference oil-based rapeseed margarine. Subsequently, the two groups will follow 2 dietary intervention periods of 3 weeks during which the volunteers will have alternatively either the reference oil/margarine or the optimized oil/margarine. Three weeks of "wash out" will separate the two dietary interventions of the cross over design trial.

Cardiovascular risk and oxidative stress biomarkers will be assessed in plasma at week 0, 3, 6, 9 and 12.

Volunteers will alsoperform dietary surveys at the week 3, 6, 9 and 12.

Post prandial study:

16 volunteers will be cast lots among the 60 volunteers. They will be randomised into 2 groups of 8. The first kinetic study will be done on week 3. 8 subjects will take 66 g of reference oil and 8 subjects will take 66 g of the optimized oil. 5 blood samples (20 mL each) will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age : 30 to 65
* Body mass index between 25 and 30 kg/m²
* Weight lower than 110 kg
* Subject considered as normal after clinical examination and medical questionnaire
* Subject giving his written informed consent
* Subject willing to comply with the study procedures
* Affiliated to National Health Insurance

Exclusion Criteria:

* Biological results judged abnormal by investigator
* Positive serologies to HIV or HCV
* Previous medical and/or surgery judged by the investigator as incompatible with the study
* Taking medicine: hypocholesterolemic,beta blockers, IEC,
* Diabetes1 and 2
* High blood pressure
* Digestive, cardiovascular, renal, liver, tumor or thyroid diseases in the last 5 years
* Infectious or inflammatory diseases in the last 5 years
* Previous heavy intestine surgery (except appendectomy)
* Triglycerides> 4 g/L
* Dyslipidemia: HDL cholesterol< 0.4 g/L or LDL/HDL>6.25
* blood donation done less than 2 month before the start of the study
* Particular diet: vegetarian, vegan...
* Anormal dietary habits
* Consumption of food complements: antioxidant, ...
* intense physical exercise practise (>5 h per week)
* Tobacco, alcohol:more than 30 g of alcohol/day, i.e.3 glasses/day, smoking > 5 cigarettes /day
* No affiliated to National Health Insurance people
* Refusal to sign informed consent
* Refusal to be registered on the National Volunteers Data file
* Currently participating or who having got 4500 E in this year before to have participated in another clinical trial

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
HDL-Cholestérol | study 1

SECONDARY OUTCOMES:
Biomarkers of the oxidative stress every 3 weeks Biomarkers of the oxidative stress during the post prandial period | every 3 weeks, during the post prandial period

CONTACTS AND LOCATIONS:
Overall Officials: Noël Cano, Principal Investigator — Centre de Recherche en Nutrition Humaine d'Auvergne
Locations (1):
- CRNH Auvergne, Clermont-Ferrand, France